CLINICAL TRIAL: NCT02951195
Title: A Phase 2, Randomized, Double Blind, Controlled Study to Evaluate the Safety of VX-152 Combination Therapy in Adults With Cystic Fibrosis
Brief Title: A Study Evaluating the Safety of VX-152 Combination Therapy in Adults With Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VX16-152-102
Record Dates: First submitted 2016-10-26; First posted 2016-11-01 (Estimated); Results first posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — tezacaftor, ivacaftor drug combination; ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Part 1: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Part 1 Cohort 1A: TC (Experimental)
  Interventions: Drug: VX-152; Drug: TEZ/IVA; Drug: IVA
- Part 1 Cohort 1B: TC (Experimental)
  Interventions: Drug: VX-152; Drug: TEZ/IVA; Drug: IVA
- Part 1 Cohort 1C: TC (Experimental)
  Interventions: Drug: VX-152; Drug: TEZ/IVA; Drug: IVA
- Part 2 Cohort 2A: TEZ/IVA (Active Comparator)
  Interventions: Drug: TEZ/IVA; Drug: IVA; Drug: Placebo
- Part 2 Cohort 2A: TC (Experimental)
  Interventions: Drug: VX-152; Drug: TEZ/IVA; Drug: IVA
- Part 2 Cohort 2B: TEZ/IVA (Active Comparator)
  Interventions: Drug: TEZ/IVA; Drug: IVA; Drug: Placebo
- Part 2 Cohort 2B: TC (Experimental)
  Interventions: Drug: VX-152; Drug: TEZ/IVA; Drug: IVA

INTERVENTIONS:
Drug: VX-152 — Tablet for oral administration.
  Arms: Part 1 Cohort 1A: TC; Part 1 Cohort 1B: TC; Part 1 Cohort 1C: TC; Part 2 Cohort 2A: TC; Part 2 Cohort 2B: TC
Drug: TEZ/IVA — Fixed-dose combination tablet for oral administration.
  Other Names: VX-661/VX-770; Tezacaftor/Ivacaftor
  Arms: Part 1 Cohort 1A: TC; Part 1 Cohort 1B: TC; Part 1 Cohort 1C: TC; Part 2 Cohort 2A: TC; Part 2 Cohort 2A: TEZ/IVA; Part 2 Cohort 2B: TC; Part 2 Cohort 2B: TEZ/IVA
Drug: IVA — Tablet for oral administration.
  Other Names: VX-770; Ivacaftor
  Arms: Part 1 Cohort 1A: TC; Part 1 Cohort 1B: TC; Part 1 Cohort 1C: TC; Part 2 Cohort 2A: TC; Part 2 Cohort 2A: TEZ/IVA; Part 2 Cohort 2B: TC; Part 2 Cohort 2B: TEZ/IVA
Drug: Placebo — Placebo matched to VX-152.
  Arms: Part 2 Cohort 2A: TEZ/IVA; Part 2 Cohort 2B: TEZ/IVA
Drug: Placebo — Placebo matched to VX-152/TEZ/IVA triple combination (TC).
  Arms: Part 1: Placebo

SUMMARY:
This is a Phase 2, randomized, double blind, placebo and active-controlled, parallel group, multicenter study designed to evaluate the safety and tolerability of VX-152 in Triple Combination (TC) with tezacaftor (TEZ; VX-661) and ivacaftor (IVA; VX-770) in subjects with cystic fibrosis (CF) who are heterozygous for the F508del mutation and a minimal function (MF) CFTR mutation not likely to respond to TEZ and/or IVA therapy (F508del/MF), or who are homozygous for the F508del mutation of the CF transmembrane conductance regulator (CFTR) gene (F508del/F508del).

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to comply with scheduled visits, treatment pan, study restrictions, laboratory tests, contraceptive guidelines, and other study procedures.
* Body weight ≥35 kg.
* Sweat chloride value ≥ 60 mmol/L from test results obtained during screening.
* Subjects must have an eligible CFTR genotype:

  * Cohorts 1A, 1B, 1C: Heterozygous for F508del and a minimal function mutation known or predicted not to respond to TEZ and/or IVA.
  * Cohorts 2A, 2B: Homozygous for F508del.
* Subjects must have an FEV1 ≥40% and ≤90% of predicted normal for age, sex, and height at the Screening Visit.
* Stable CF disease as judged by the investigator.
* Willing to remain on a stable CF medication regimen through the planned end of treatment or if applicable the Safety Follow-up Visit.

Exclusion Criteria:

* History of any comorbidity that in the opinion of the investigator might confound the results of the study or pose an additional risk in administering study drug to the subject.
* History of cirrhosis with portal hypertension.
* Risk factors for Torsade de Pointes.
* History of hemolysis.
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency assessed at Screening.
* Clinically significant abnormal laboratory values at screening.
* An acute upper or lower respiratory infection, pulmonary exacerbation, or changes in therapy for pulmonary disease within 28 days before the first dose of study drug.
* Lung infection with organisms associated with a more rapid decline in pulmonary status.
* An acute illness not related to CF within 14 days before the first dose of study drug.
* A standard digital ECG demonstrating QTc >450 msec at screening.
* History of solid organ or hematological transplantation.
* History or evidence of cataract or lens opacity determined to be clinically significant by the ophthalmologist or optometrist, based on the ophthalmologic examination during the Screening Period.
* History of alcohol or drug abuse in the past year, including but not limited to, cannabis, cocaine, and opiates, as deemed by the investigator.
* Ongoing or prior participation in an investigational drug study with certain exceptions.
* Use of commercially available CFTR modulator within 14 days before screening (applies only to Cohorts 1A, 1B, and 1C).
* Pregnant or nursing females: Females of childbearing potential must have a negative pregnancy test at screening and Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Birmingham, Alabama
  - La Jolla, California
  - Los Angeles, California
  - Orlando, Florida
  - Chicago, Illinois
  - Peoria, Illinois
  - St Louis, Missouri
  - Chapel Hill, North Carolina
  - Akron, Ohio
  - Cleveland, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Fort Worth, Texas
  - Houston, Texas
  - Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 80 participants were enrolled in the study (34 participants in Part 1 and 46 participants in Part 2). Out of 46 participants enrolled in Part 2, 4 participants discontinued during the run-in period and were not randomized in the treatment period. Therefore, results are presented for 76 participants in this study.
Groups:
- Part 1: Placebo: Participants received placebo matched to VX-152/TEZ/IVA triple combination (TC) for 2 weeks.
- Part 1 Cohort 1A: TC: Participants received VX-152 100 milligram (mg) every 12 hours (q12h)/TEZ 100 mg once daily (qd)/IVA 150 mg q12h TC for 2 weeks.
- Part 1 Cohort 1B: TC: Participants received VX-152 200 mg q12h/TEZ 100 mg qd/IVA 150 mg q12h TC for 2 weeks.
- Part 1 Cohort 1C: TC: Participants received VX-152 300 mg q12h/TEZ 100 mg qd/IVA 150 mg q12h TC for 2 weeks.
- Part 2 Cohort 2A: TEZ/IVA: Following run-in period on TEZ 100 mg qd/IVA 150 mg q12h for 4 weeks, participants received placebo matched to VX-152 and TEZ 100 mg qd/IVA 150 mg q12h for 2 weeks in treatment period and TEZ 100 mg qd/IVA 150 mg q12h for 2 weeks in washout period.
- Part 2 Cohort 2A: TC: Following run-in period on TEZ 100 mg qd/IVA 150 mg q12h for 4 weeks, participants received VX-152 200 mg q12h/TEZ 100 mg qd/IVA 150 mg q12h TC for 2 weeks in treatment period and TEZ 100 mg qd/IVA 150 mg q12h for 2 weeks in washout period.
- Part 2 Cohort 2B: TEZ/IVA: Following run-in period on TEZ 100 mg qd/IVA 150 mg q12h for 4 weeks, participants received placebo matched to VX-152 and TEZ 100 mg qd/IVA 150 mg q12h for 4 weeks in treatment period and TEZ 100 mg qd/IVA 150 mg q12h for 2 weeks in washout period.
- Part 2 Cohort 2B: TC: Following run-in period on TEZ 100 mg qd/IVA 150 mg q12h for 4 weeks, participants received VX-152 300 mg q12h/TEZ 100 mg qd/IVA 150 mg q12h TC for 4 weeks in treatment period and TEZ 100 mg qd/IVA 150 mg q12h for 2 weeks in washout period.
Period: Overall Study
Arm/Group | Part 1: Placebo | Part 1 Cohort 1A: TC | Part 1 Cohort 1B: TC | Part 1 Cohort 1C: TC | Part 2 Cohort 2A: TEZ/IVA | Part 2 Cohort 2A: TC | Part 2 Cohort 2B: TEZ/IVA | Part 2 Cohort 2B: TC
Started | 8 | 6 | 10 | 10 | 4 | 10 | 7 | 21
Completed | 8 | 6 | 10 | 10 | 4 | 10 | 7 | 21
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1: Placebo: Participants received placebo matched to VX-152/TEZ/IVA TC for 2 weeks.
- Part 1 Cohort 1A: TC: Participants received VX-152 100 mg q12h/TEZ 100 mg qd/IVA 150 mg q12h TC for 2 weeks.
- Total: Total of all reporting groups
Arm/Group | Part 1: Placebo | Part 1 Cohort 1A: TC | Part 1 Cohort 1B: TC | Part 1 Cohort 1C: TC | Part 2 Cohort 2A: TEZ/IVA | Part 2 Cohort 2A: TC | Part 2 Cohort 2B: TEZ/IVA | Part 2 Cohort 2B: TC | Total
Number analyzed (Participants) | 8 | 6 | 10 | 10 | 4 | 10 | 7 | 21 | 76
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=18 and <65 years | 8 | 6 | 10 | 10 | 4 | 10 | 7 | 21 | 76
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 4 | 3 | 2 | 6 | 4 | 14 | 39
  Male | 4 | 4 | 6 | 7 | 2 | 4 | 3 | 7 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
  Not Hispanic or Latino | 6 | 6 | 10 | 9 | 4 | 10 | 7 | 21 | 73
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 7 | 5 | 10 | 10 | 4 | 10 | 7 | 21 | 74
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) [Count of Participants; unit: Participants] — FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
  Participants
    <40 percent | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 4
    ≥40 to <70 percent | 5 | 6 | 7 | 4 | 3 | 10 | 5 | 18 | 58
    ≥70 to ≤90 percent | 2 | 0 | 1 | 5 | 1 | 0 | 2 | 3 | 14
    >90 percent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability as Assessed by Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 Through Safety Follow-up Visit (Up to Day 43 for Part 1 and Day 71 for Part 2)
Population: Safety Set included all participants who received at least 1 dose of study drug in the treatment period.
Measure: Number; unit: participants
Arm/Group | Part 1: Placebo | Part 1 Cohort 1A: TC | Part 1 Cohort 1B: TC | Part 1 Cohort 1C: TC | Part 2 Cohort 2A: TEZ/IVA | Part 2 Cohort 2A: TC | Part 2 Cohort 2B: TEZ/IVA | Part 2 Cohort 2B: TC
Number analyzed (Participants) | 8 | 6 | 10 | 10 | 4 | 10 | 7 | 21
participants
  Participants with TEAEs | 8 | 3 | 7 | 10 | 3 | 6 | 5 | 19
  Participants with SAEs | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0

2. Primary Outcome: Absolute Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) at Day 15 for Part 1 and Part 2 Cohort 2A
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline at Day 15
Population: Full Analysis Set (FAS) included all randomized participants with the intended cystic fibrosis transmembrane conductance regulator protein (CFTR) allele mutation who received at least 1 dose of study drug in the treatment period. As pre-specified in analysis plan, only Part 1 and Part 2 Cohort 2A arms were assessed for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage points
Arm/Group | Part 1: Placebo | Part 1 Cohort 1A: TC | Part 1 Cohort 1B: TC | Part 1 Cohort 1C: TC | Part 2 Cohort 2A: TEZ/IVA | Part 2 Cohort 2A: TC
Number analyzed (Participants) | 8 | 6 | 10 | 10 | 4 | 10
percentage points | -0.8 [-4.8 to 3.3] | 5.7 [1.0 to 10.3] | 9.7 [6.1 to 13.3] | 8.0 [4.0 to 12.0] | -1.0 [-9.9 to 7.8] | 7.3 [1.9 to 12.6]
Statistical Analysis 1: Comparison: Part 1: Placebo vs Part 1 Cohort 1A: TC; Test type: Superiority; p = 0.0207, Mixed-effects Model for Repeated Measure; LS Mean Difference = 6.4, 95% CI 2-sided [0.3 to 12.6]
Statistical Analysis 2: Comparison: Part 1: Placebo vs Part 1 Cohort 1B: TC; Test type: Superiority; p = 0.0002, Mixed-effects Model for Repeated Measure; LS Mean Difference = 10.5, 95% CI 2-sided [5.0 to 15.9]
Statistical Analysis 3: Comparison: Part 1: Placebo vs Part 1 Cohort 1C: TC; Test type: Superiority; p = 0.0019, Mixed-effects Model for Repeated Measure; LS Mean Difference = 8.8, 95% CI 2-sided [3.0 to 14.5]
Statistical Analysis 4: Comparison: Part 2 Cohort 2A: TEZ/IVA vs Part 2 Cohort 2A: TC; Test type: Superiority; p = 0.0540, Mixed-effects Model for Repeated Measure; LS Mean Difference = 8.3, 95% CI 2-sided [-2.1 to 18.7]

3. Primary Outcome: Absolute Change in ppFEV1 Through Day 29 for Part 2 Cohort 2B
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline Through Day 29
Population: FAS. As pre-specified in analysis plan, only Part 2 Cohort 2B arms were assessed for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage points
Arm/Group | Part 2 Cohort 2B: TEZ/IVA | Part 2 Cohort 2B: TC
Number analyzed (Participants) | 7 | 21
percentage points | -2.2 [-6.6 to 2.1] | 6.5 [4.0 to 9.0]
Statistical Analysis 1: Comparison: Part 2 Cohort 2B: TEZ/IVA vs Part 2 Cohort 2B: TC; Test type: Superiority; p = 0.0007, Mixed-effects Model for Repeated Measure; LS Mean Difference = 8.7, 95% CI 2-sided [3.7 to 13.8]

4. Secondary Outcome: Absolute Change in Sweat Chloride Concentrations at Day 15 for Part 1 and Part 2 Cohort 2A
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline at Day 15
Population: FAS. As pre-specified in analysis plan, only Part 1 and Part 2 Cohort 2A arms were assessed for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimole per liter (mmol/L)
Arm/Group | Part 1: Placebo | Part 1 Cohort 1A: TC | Part 1 Cohort 1B: TC | Part 1 Cohort 1C: TC | Part 2 Cohort 2A: TEZ/IVA | Part 2 Cohort 2A: TC
Number analyzed (Participants) | 8 | 6 | 10 | 10 | 4 | 10
millimole per liter (mmol/L) | -0.1 [-8.4 to 8.3] | -19.5 [-29.1 to -10.0] | -13.6 [-21.4 to -5.8] | -27.5 [-35.0 to -20.1] | 3.5 [-9.2 to 16.2] | -21.3 [-29.5 to -13.1]
Statistical Analysis 1: Comparison: Part 1: Placebo vs Part 1 Cohort 1A: TC; Test type: Superiority; p = 0.0018, Mixed-effects Model for Repeated Measure; Least Squares (LS) Mean Difference = -19.5, 95% CI 2-sided [-32.2 to -6.8]
Statistical Analysis 2: Comparison: Part 1: Placebo vs Part 1 Cohort 1B: TC; Test type: Superiority; p = 0.0106, Mixed-effects Model for Repeated Measure; LS Mean Difference = -13.6, 95% CI 2-sided [-25.0 to -2.1]
Statistical Analysis 3: Comparison: Part 1: Placebo vs Part 1 Cohort 1C: TC; Test type: Superiority; p < 0.0001, Mixed-effects Model for Repeated Measure; LS Mean Difference = -27.5, 95% CI 2-sided [-38.6 to -16.3]
Statistical Analysis 4: Comparison: Part 2 Cohort 2A: TEZ/IVA vs Part 2 Cohort 2A: TC; Test type: Superiority; p = 0.0017, Mixed-effects Model for Repeated Measure; LS Mean Difference = -24.8, 95% CI 2-sided [-40.0 to -9.7]

5. Secondary Outcome: Absolute Change in Sweat Chloride Concentrations Through Day 29 for Part 2 Cohort 2B
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline Through Day 29
Population: FAS. As pre-specified in analysis plan, only Part 2 Cohort 2B arms were assessed for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Part 2 Cohort 2B: TEZ/IVA | Part 2 Cohort 2B: TC
Number analyzed (Participants) | 7 | 21
mmol/L | 1.6 [-6.8 to 10.0] | -22.3 [-27.3 to -17.3]
Statistical Analysis 1: Comparison: Part 2 Cohort 2B: TEZ/IVA vs Part 2 Cohort 2B: TC; Test type: Superiority; p < 0.0001, Mixed-effects Model for Repeated Measure; LS Mean Difference = -23.9, 95% CI 2-sided [-33.7 to -14.1]

6. Secondary Outcome: Relative Change in ppFEV1 at Day 15 for Part 1 and Part 2 Cohort 2A
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline at Day 15
Population: FAS. As pre-specified in analysis plan, only Part 1 and Part 2 Cohort 2A arms were assessed for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Groups:
- Part 1: Placebo: Participants received placebo matched to VX-152/TEZ/IVA for 2 weeks.
Arm/Group | Part 1: Placebo | Part 1 Cohort 1A: TC | Part 1 Cohort 1B: TC | Part 1 Cohort 1C: TC | Part 2 Cohort 2A: TEZ/IVA | Part 2 Cohort 2A: TC
Number analyzed (Participants) | 8 | 6 | 10 | 10 | 4 | 10
percent change | -2.3 [-9.8 to 5.3] | 10.3 [1.6 to 19.0] | 19.0 [12.3 to 25.8] | 14.8 [7.3 to 22.4] | -1.4 [-17.1 to 14.4] | 13.2 [3.7 to 22.7]
Statistical Analysis 1: Comparison: Part 1: Placebo vs Part 1 Cohort 1A: TC; Test type: Superiority; p = 0.0166, Mixed-effects Model for Repeated Measure; LS Mean Difference = 12.5, 95% CI 2-sided [1.1 to 24.0]
Statistical Analysis 2: Comparison: Part 1: Placebo vs Part 1 Cohort 1B: TC; Test type: Superiority; p < 0.0001, Mixed-effects Model for Repeated Measure; LS Mean Difference = 21.3, 95% CI 2-sided [11.2 to 31.4]
Statistical Analysis 3: Comparison: Part 1: Placebo vs Part 1 Cohort 1C: TC; Test type: Superiority; p = 0.0013, Mixed-effects Model for Repeated Measure; LS Mean Difference = 17.1, 95% CI 2-sided [6.3 to 27.8]
Statistical Analysis 4: Comparison: Part 2 Cohort 2A: TEZ/IVA vs Part 2 Cohort 2A: TC; Test type: Superiority; p = 0.0563, Mixed-effects Model for Repeated Measure; LS Mean Difference = 14.5, 95% CI 2-sided [-3.8 to 32.9]

7. Secondary Outcome: Relative Change in ppFEV1 Through Day 29 for Part 2 Cohort 2B
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline Through Day 29
Population: FAS. As pre-specified in analysis plan, only Part 2 Cohort 2B arms were assessed for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Part 2 Cohort 2B: TEZ/IVA | Part 2 Cohort 2B: TC
Number analyzed (Participants) | 7 | 21
percent change | -2.0 [-9.2 to 5.1] | 11.5 [7.4 to 15.7]
Statistical Analysis 1: Comparison: Part 2 Cohort 2B: TEZ/IVA vs Part 2 Cohort 2B: TC; Test type: Superiority; p = 0.0012, Mixed-effects Model for Repeated Measure; LS Mean Difference = 13.6, 95% CI 2-sided [5.3 to 21.9]

8. Secondary Outcome: Absolute Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score at Day 15 for Part 1 and Part 2 Cohort 2A
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms, score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life.
Time Frame: From Baseline at Day 15
Population: FAS. As pre-specified in analysis plan, only Part 1 and Part 2 Cohort 2A arms were assessed for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Part 1: Placebo | Part 1 Cohort 1A: TC | Part 1 Cohort 1B: TC | Part 1 Cohort 1C: TC | Part 2 Cohort 2A: TEZ/IVA | Part 2 Cohort 2A: TC
Number analyzed (Participants) | 8 | 6 | 10 | 10 | 4 | 10
units on a scale | -7.6 [-18.6 to 3.4] | 6.6 [-6.0 to 19.1] | 21.8 [12.1 to 31.6] | 18.6 [8.8 to 28.5] | 5.8 [-8.0 to 19.6] | 10.6 [1.9 to 19.2]
Statistical Analysis 1: Comparison: Part 1: Placebo vs Part 1 Cohort 1A: TC; Test type: Superiority; p = 0.0476, ANCOVA; LS Mean Difference = 14.1, 95% CI 2-sided [-2.6 to 30.9]
Statistical Analysis 2: Comparison: Part 1: Placebo vs Part 1 Cohort 1B: TC; Test type: Superiority; p = 0.0001, ANCOVA; LS Mean Difference = 29.4, 95% CI 2-sided [14.8 to 44.0]
Statistical Analysis 3: Comparison: Part 1: Placebo vs Part 1 Cohort 1C: TC; Test type: Superiority; p = 0.0006, ANCOVA; LS Mean Difference = 26.2, 95% CI 2-sided [11.3 to 41.1]
Statistical Analysis 4: Comparison: Part 2 Cohort 2A: TEZ/IVA vs Part 2 Cohort 2A: TC; Test type: Superiority; p = 0.2714, Mixed-effects Model for Repeated Measure; LS Mean Difference = 4.8, 95% CI 2-sided [-11.6 to 21.2]

9. Secondary Outcome: Absolute Change From Baseline in CFQ-R Respiratory Domain Score at Day 29 for Part 2 Cohort 2B
Description: as for outcome 8
Time Frame: From Baseline at Day 29
Population: FAS. As pre-specified in analysis plan, only Part 2 Cohort 2B arms were assessed for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Part 2 Cohort 2B: TEZ/IVA | Part 2 Cohort 2B: TC
Number analyzed (Participants) | 7 | 21
units on a scale | 4.8 [-3.7 to 13.3] | 16.1 [11.2 to 21.0]
Statistical Analysis 1: Comparison: Part 2 Cohort 2B: TEZ/IVA vs Part 2 Cohort 2B: TC; Test type: Superiority; p = 0.0138, Mixed-effects Model for Repeated Measure; LS Mean Difference = 11.3, 95% CI 2-sided [1.3 to 21.2]

10. Secondary Outcome: Pre-dose Plasma Concentration (Ctrough) of VX-152, TEZ, M1-TEZ, IVA, and M1-IVA
Time Frame: Pre-dose at Day 8, Day 15 and Day 29
Population: Pharmacokinetic Set (PK) included all participants who received at least 1 dose of study drug in treatment period. Here "Number Analyzed" signifies those participants who were evaluable at specified time points. Day 29 assessments were planned for Part 2: Cohort 2B groups only. VX-152 Ctrough category was not applicable to Part 2: TEZ/IVA groups.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- Part 1 Cohort 1A: TC: Participants received VX-152 100 mg q12h/TEZ 100 qd/IVA 150 mg q12h TC for 2 weeks.
Arm/Group | Part 1 Cohort 1A: TC | Part 1 Cohort 1B: TC | Part 1 Cohort 1C: TC | Part 2 Cohort 2A: TEZ/IVA | Part 2 Cohort 2A: TC | Part 2 Cohort 2B: TEZ/IVA | Part 2 Cohort 2B: TC
Number analyzed (Participants) | 6 | 10 | 10 | 4 | 10 | 7 | 21
nanogram per milliliter (ng/mL)
  Day 8: VX-152: number analyzed (Participants) | 6 | 10 | 10 | 0 | 10 | 0 | 21
  Day 8: VX-152 | 167 (65.4) | 240 (370) | 538 (576) |  | 355 (287) |  | 463 (730)
  Day 15: VX-152: number analyzed (Participants) | 6 | 10 | 10 | 0 | 9 | 0 | 20
  Day 15: VX-152 | 173 (72.1) | 278 (212) | 804 (812) |  | 554 (429) |  | 560 (657)
  Day 29: VX-152: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 17
  Day 29: VX-152 |  |  |  |  |  |  | 698 (1040)
  Day 8: TEZ | 2610 (1400) | 1500 (1140) | 1680 (996) | 1900 (1730) | 1830 (693) | 2010 (669) | 1460 (1470)
  Day 15: TEZ: number analyzed (Participants) | 6 | 10 | 10 | 4 | 9 | 7 | 20
  Day 15: TEZ | 2450 (2000) | 1220 (545) | 1180 (495) | 1120 (135) | 1620 (1030) | 1970 (1040) | 1050 (543)
  Day 29: TEZ: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 6 | 17
  Day 29: TEZ |  |  |  |  |  | 2470 (1060) | 1190 (422)
  Day 8: M1-TEZ | 4520 (1090) | 3060 (1480) | 3490 (1640) | 3760 (1100) | 4900 (1050) | 4980 (1450) | 4150 (1280)
  Day 15: M1-TEZ: number analyzed (Participants) | 6 | 10 | 9 | 4 | 9 | 7 | 20
  Day 15: M1-TEZ | 4680 (1020) | 2890 (898) | 3310 (1220) | 3430 (824) | 4270 (1280) | 4420 (1810) | 3650 (1320)
  Day 29: M1-TEZ: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 6 | 17
  Day 29: M1-TEZ |  |  |  |  |  | 4280 (1650) | 3680 (742)
  Day 8: IVA | 779 (442) | 522 (401) | 545 (234) | 702 (425) | 610 (262) | 953 (360) | 434 (251)
  Day 15: IVA: number analyzed (Participants) | 6 | 10 | 10 | 4 | 9 | 7 | 20
  Day 15: IVA | 841 (588) | 535 (310) | 467 (236) | 441 (300) | 645 (373) | 863 (488) | 389 (222)
  Day 29: IVA: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 6 | 17
  Day 29: IVA |  |  |  |  |  | 1010 (446) | 468 (279)
  Day 8: M1-IVA | 1590 (1050) | 1040 (947) | 1330 (747) | 1660 (1200) | 1470 (671) | 1810 (665) | 1170 (551)
  Day 15: M1-IVA: number analyzed (Participants) | 6 | 10 | 9 | 4 | 9 | 7 | 20
  Day 15: M1-IVA | 1230 (326) | 1200 (848) | 1140 (550) | 1030 (762) | 1510 (891) | 1620 (760) | 1100 (598)
  Day 29: M1-IVA: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 6 | 17
  Day 29: M1-IVA |  |  |  |  |  | 1890 (659) | 1240 (705)

ADVERSE EVENTS:
Time Frame: Day 1 Through Safety Follow-up Visit (Up to Day 43 for Part 1 and Day 71 for Part 2)
Arm/Group | Part 1: Placebo | Part 1 Cohort 1A: TC | Part 1 Cohort 1B: TC | Part 1 Cohort 1C: TC | Part 2 Cohort 2A: TEZ/IVA | Part 2 Cohort 2A: TC | Part 2 Cohort 2B: TEZ/IVA | Part 2 Cohort 2B: TC
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/10 | 0/10 | 0/4 | 0/10 | 0/7 | 0/21
Serious Adverse Events (participants affected / at risk) | 2/8 | 0/6 | 0/10 | 1/10 | 0/4 | 0/10 | 0/7 | 0/21
Other Adverse Events (participants affected / at risk) | 8/8 | 3/6 | 7/10 | 9/10 | 3/4 | 6/10 | 5/7 | 18/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo (N=8) | Part 1 Cohort 1A: TC (N=6) | Part 1 Cohort 1B: TC (N=10) | Part 1 Cohort 1C: TC (N=10) | Part 2 Cohort 2A: TEZ/IVA (N=4) | Part 2 Cohort 2A: TC (N=10) | Part 2 Cohort 2B: TEZ/IVA (N=7) | Part 2 Cohort 2B: TC (N=21)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo (N=8) | Part 1 Cohort 1A: TC (N=6) | Part 1 Cohort 1B: TC (N=10) | Part 1 Cohort 1C: TC (N=10) | Part 2 Cohort 2A: TEZ/IVA (N=4) | Part 2 Cohort 2A: TC (N=10) | Part 2 Cohort 2B: TEZ/IVA (N=7) | Part 2 Cohort 2B: TC (N=21)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Post-tussive vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Thirst (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vessel puncture site haemorrhage (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 3 | 0 | 1 | 0 | 0 | 1 | 3 | 5
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Procedural dizziness (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Platelet count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 3 | 1 | 0 | 0 | 4
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4
Breast discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breast tenderness (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 1 | 1 | 1 | 0 | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 2
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 2 | 0 | 0 | 0 | 3
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 2
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 1 | 0 | 1 | 1 | 6
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-04-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT02951195/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-27): https://cdn.clinicaltrials.gov/large-docs/95/NCT02951195/SAP_001.pdf